CLINICAL TRIAL: NCT02331303
Title: A Drug Utilization Study of Xofigo Use in Sweden
Brief Title: A Drug Utilization Study of Radium-223 in Sweden
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17399
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group1: This is a single-arm descriptive observational drug utilization study based on secondary data collection of patients treated with Xofigo in Sweden.
  This study will include patients receiving treatment of Xofigo at certified nuclear medicine centers across Sweden during a two year period.
  Interventions: Other: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Other: Radium-223 dichloride (Xofigo, BAY88-8223) — Xofigo was approved in the US and EU for the following indication: Xofigo is indicated for the treatment of adults with castration-resistant prostate cancer, symptomatic bone metastases and no known visceral metastases. Xofigo is contraindicated in women who are or may become pregnant.

SUMMARY:
The objective of this study is to evaluate the extent of potential off-label use of Xofigo in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving Xofigo with data recorded at nuclear medicine centers in Sweden between 01 July 2014 and 30 June 2016 will be included in the study

Exclusion Criteria:

* Patients receiving Xofigo in a clinical trial will not be included in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include patients receiving treatment of Xofigo at certified nuclear medicine centers across Sweden during a two year period. It will consist of mCRPC patients and potentially some other patient groups in whom Xofigo may be used off-label including women, children, cancer patients having bone metastasis with a diagnosis other than CRPC, and patients with repeated courses of treatment or in excess of those recommended in the label. This study will be based on data extracted from two pre-established data sources: 15 nuclear medicine centers across Sweden and the Swedish National Cancer Registry.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Proportion of men with metastatic castration resistant prostate cancer (mCRPC) of Xofigo use | Up to 2 years
Proportion of being women of Xofigo use | Up to 2 years
Proportion of being children of Xofigo use | Up to 2 years
Proportion of bone metastasis but having a diagnosis of other cancer than mCRPV | Up to 2 years
Dosage of Xofigo (kBq/kg) | Up to 2 years
Proportion of participants of dose outside label recommendation | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Stockholm, Sweden